CLINICAL TRIAL: NCT03936998
Title: VE416 and Low-dose Peanut Oral Immunotherapy for Treatment of Persistent Peanut Allergy
Brief Title: VE416 for Treatment of Food Allergy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Vedanta Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Wayne G. Shreffler, MD, PhD, Director of the Food Allergy Center, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P000886
Record Dates: First submitted 2019-04-17; First posted 2019-05-03 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, double-blind trial with four arms evaluating VE416 as pretreatment or concurrent treatment in comparison to low-dose peanut oral immunotherapy (PNOIT) alone.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- vancomycin plus VE416 before PNOIT (Experimental): active vancomycin plus VE416 before PNOIT
  Interventions: Combination Product: Vancomycin plus VE416 before PNOIT
- Vancomycin plus VE416 with PNOIT (Experimental): active vancomycin plus active VE416 with active PNOIT
  Interventions: Combination Product: Vancomycin plus VE416 with PNOIT
- Placebo plus VE416 with PNOIT (Experimental): placebo vancomycin plus active VE416 with active VE416
  Interventions: Combination Product: Placebo plus VE416 with PNOIT
- Placebo plus placebo with PNOIT (Active Comparator): placebo vancomycin and placebo VE416 with active peanut oral immunotherapy
  Interventions: Combination Product: Placebo plus placebo with PNOIT

INTERVENTIONS:
Combination Product: Vancomycin plus VE416 before PNOIT — Vancomycin PO QD x 5 days, followed by VE416 PO QD x 6 weeks followed by PNOIT
  Arms: vancomycin plus VE416 before PNOIT
Combination Product: Vancomycin plus VE416 with PNOIT — Placebo for vancomycin for 5 days and placebo for VE416 x 6 weeks, followed by Vancomycin PO QD x 5 days, followed by VE416 PO QD x 6 weeks with concomitant PNOIT
  Arms: Vancomycin plus VE416 with PNOIT
Combination Product: Placebo plus VE416 with PNOIT — Placebo for vancomycin for 5 days and placebo for VE416 x 6 weeks, followed by placebo for vancomycin PO QD x 5 days, followed by VE416 PO QD x 6 weeks with concomitant PNOIT
  Arms: Placebo plus VE416 with PNOIT
Combination Product: Placebo plus placebo with PNOIT — Placebo for vancomycin for 5 days and placebo for VE416 x 6 weeks, followed by placebo for vancomycin PO QD x 5 days, followed by placebo for VE416 PO QD x 6 weeks with concomitant PNOIT
  Arms: Placebo plus placebo with PNOIT

SUMMARY:
This is a single-center, randomized, double-blind trial with four arms evaluating VE416 as pretreatment or concurrent treatment in comparison to low-dose peanut oral immunotherapy (PNOIT) alone.

DETAILED DESCRIPTION:
In this research study the investigators want to learn more about an investigational medicine called VE416 in combination with vancomycin (an antibiotic) while undergoing peanut oral immunotherapy. VE416 is a combination of dormant (inactive) bacteria given in a capsule. The bacteria are reactivated once they reach participants intestines and in combination with peanut flour may help to prevent participants from getting sick (upset stomach, breathing problems, and skin problems) when participants come into contact with peanuts.

The investigators are doing this research study to find out if VE416 in combination with vancomycin (an antibiotic) while undergoing peanut oral immunotherapy can help people with peanut allergy. VE416 is a consortium of commensal, or "friendly", dormant (inactive) bacteria given in a capsule. The bacteria are reactivated once they reach participants intestines. The investigators also want to find out if VE416 with peanut oral immunotherapy is safe to take without causing too many side effects.

ELIGIBILITY:
Inclusion Criteria:

* People of all ethnic/racial/gender groups aged 12-55 years old with a documented medical history of peanut allergy.
* Evidence of peanut-specific IgE by either: positive skin prick test to peanut (reaction wheal at least 5 mm larger than saline control) or serum peanut-specific IgE _5 kU/L at screening visit.
* Ara h 2 specific IgE >0.35 kU/L at screening visit.
* Willing to sign informed consent or whose parent or legal guardian is willing to sign the consent form (age appropriate).
* Willing to sign the assent form, if age appropriate.
* (For continuation into Phase II only) Allergic reaction requiring treatment at _ 100 mg dose of peanut protein during Entry Challenge.

Exclusion Criteria:

* History of severe anaphylaxis as defined by hypoxia (cyanosis or SpO2 <92% during reaction), documented hypotension (documented systolic BP >30% below predicted normal for sex, height, weight or from known baseline), neurological compromise (confusion, loss of consciousness), or incontinence.
* Severe or Moderate asthma as defined using the severity criteria of the current NHLBI Guidelines for the Diagnosis and Management of Asthma (http://www.nhlbi.nih.gov/guidelines/asthma/).
* Poorly-controlled asthma as defined by FEV1 <80% or any of the following symptoms: nighttime awakening >2 days/week or rescue medication use >2 days / week.
* Diagnosis of other severe or complicating medical problems, including autoimmune or chronic immune inflammatory conditions or gastrointestinal inflammatory conditions, including Celiac Disease, Inflammatory Bowel Disease and Eosinophilic Gastrointestinal Disorders
* Inability to cooperate with and/or perform oral food challenge procedures.
* Inability to swallow size 0 capsule
* Primary Immune Deficiency
* Allergy to oat confirmed by skin prick testing and history
* Current use of beta blockers, angiotensin converting enzyme inhibitors, or monoamine oxidase inhibitors
* Women of childbearing potential who are pregnant, planning to become pregnant, or breastfeeding
* Hematocrit <0.36 for adult females or <0.38 for adult males Weight <23 kg
* Use within the past 6 months of other systemic immunomodulatory treatments including allergen immunotherapy, or use of biologics with an immune target, including omalizumab.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study may also exclude a participant from the study.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint- Phase 1b | 7 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Primary Endpoint- Phase II | 23 weeks, with 24 week Post-Phase II maintenance phase followed by a DBPCFC
  The geometric mean of the maximum tolerated dose (MTD) of peanut protein at DBPCFC1

SECONDARY OUTCOMES:
Secondary Endpoint- Efficacy | 54 weeks
  The percentage of patients tolerating 600 mg (1030 mg cumulative) at DBPCFC1 without treatment
Secondary Endpoint- Safety | 54 weeks
  The occurrence of treatment related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wayne G Shreffler, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berin MC. Dysbiosis in food allergy and implications for microbial therapeutics. J Clin Invest. 2021 Jan 19;131(2):e144994. doi: 10.1172/JCI144994. PMID 33463542